CLINICAL TRIAL: NCT05457608
Title: Clinical Evaluation of Clariti Monthly Multifocal and Clariti 1 Day Multifocal
Brief Title: Clinical Evaluation of Two Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-136
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2022-09

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: All participants received Lens A and then Lens B in fixed-sequence order.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A (Experimental): All participants wore lens A for 15 minutes (Period 1)
  Interventions: Device: Lens A
- Lens B (Experimental): All participants wore lens B for 15 minutes (Period 2)
  Interventions: Device: Lens B

INTERVENTIONS:
Device: Lens A — monthly replacement multifocal silicone hydrogel contact lens 15 minutes of daily wear
  Arms: Lens A
Device: Lens B — daily disposable multifocal silicone hydrogel contact lens 15 minutes of daily wear
  Arms: Lens B

SUMMARY:
The aim of this study is to evaluate the patient subjective experiences of the monthly multifocal lens when compared to the daily disposable multifocal lens after 15 minutes of daily wear.

DETAILED DESCRIPTION:
This is a single-blind, interventional, prospective, direct refit, bilateral wear study.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 42 years of age and has full legal capacity to volunteer.
* Has read and signed an information consent letter.
* Self-reports having a full eye examination in the previous two years.
* Anticipates being able to wear the study lenses for at least 8 hours a day, 5 days a week.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Habitually wears multifocal soft contact lenses, or sphere lenses for monovision, or sphere lenses for monovision, or sphere lenses for distance vision correction and use spectacles for near vision correction, for the past 3 months minimum.
* Has refractive astigmatism no higher than -0.75DC.
* Is presbyopic and requires a reading addition of at least +0.75D and no more than +2.50D.
* Can be fit and achieve binocular distance vision of at least 20/30 Snellen (or +0.20 logMAR) which participants also deem to be 'acceptable', with the available study lens parameters (powers +4.00 to -6.00DS).

Exclusion Criteria:

* Is participating in any concurrent clinical or research study.
* Has any known active ocular disease and/or infection that contraindicates contact lens wear.
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable.
* Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable.
* Has known sensitivity to the diagnostic sodium fluorescein used in the study.
* Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment.
* Has undergone refractive error surgery or intraocular surgery.

Min Age: 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-06-25 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2022-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubén V Guerrero, MSc, FIACLE, Principal Investigator — School of Optometry, National Autonomous University (UNAM)
Locations (1):
- School of Optometry Clinic, National Autonomous University (UNAM), Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-two participants were screened. All participants wore Lens A first for 15 minutes and then wore Lens B for 15 minutes.
  All the participants who were in the study were included in the analysis. (n=42)
Groups:
- Lens A: All participants wore Lens A for 15 minutes. (Period 1)
- Lens B: All participants wore Lens B for 15 minutes. (Period 2)
Period: Period 1: Lens A (15 Minutes)
Arm/Group | Lens A | Lens B
Started | 42 | 0 (All participants received Lens A in Period 1.)
Completed | 42 | 0
Not Completed | 0 | 0
Period: Period 2: Lens B (15 Minutes)
Arm/Group | Lens A | Lens B
Started | 0 (All participants received Lens B in Period 2.) | 42
Completed | 0 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall study
Groups:
- All Study Participants: Includes all study participants.
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  Lens A: <=18 years | 0
  Lens A: Between 18 and 65 years | 42
  Lens A: >=65 years | 0
  Lens B: <=18 years | 0
  Lens B: Between 18 and 65 years | 42
  Lens B: >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Comfort Ratings on Insertion
Description: Subjective comfort ratings on insertion were measured on a scale from 0 - 10, where 0= extremely uncomfortable and 10= can't feel.
Time Frame: At insertion
Population: [Not Specified]
Measure: Mean (Standard Deviation); unit: Units on scale
Groups:
- Lens A: Participants that received Lens A.
- Lens B: Participants that received Lens B.
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 42 | 42
Units on scale | 9.19 (0.86) | 9.47 (0.67)

ADVERSE EVENTS:
Time Frame: From dispense up to 15 minutes on each lens type
Description: [Not Specified]
Groups:
- Lens A: Participants wore Lens A for 15 minutes.
- Lens B: Participants wore Lens B for 15 minutes.
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT05457608/Prot_SAP_000.pdf